CLINICAL TRIAL: NCT06523530
Title: Effect of the Pharmacological Cessation of Menstruation With a GnRH Analog on Hepatic Steatosis in Women With Endometriosis
Brief Title: Effect of a GnRH Analog on Hepatic Steatosis
Acronym: EndomMASLD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Stergios A Polyzos, Associate Professor of Pharmacology, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5221
Record Dates: First submitted 2024-07-10; First posted 2024-07-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Nonalcoholic Fatty Liver; Endometriosis
Keywords: endometriosis; goserelin acetate; hepatic fibrosis; MASLD; MASH; metabolic dysfunction-associated steatotic liver disease; metabolic dysfunction-associated steatohepatitis; NAFLD; NASH; nonalcoholic fatty liver disease; nonalcoholic steatohepatitis; treatment; menopause
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Endometriosis; Liver Cirrhosis | interventions — Goserelin; Drug Implants

STUDY DESIGN:
Intervention Model Description: Multicenter, interventional, open label, non-randomized, parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Goserelin (Experimental): 31 women with histologically confirmed endometriosis will receive goserelin acetate post-surgically.
  Interventions: Drug: Goserelin Acetate 3.6 mg inj, implant
- Control (No Intervention): 31 women with histologically confirmed endometriosis will not receive pharmacological treatment post-surgically.

INTERVENTIONS:
Drug: Goserelin Acetate 3.6 mg inj, implant — 3.6 mg (1ml) administered subcutaneously once every month for 6 months (totally 6 injections)
  Other Names: Zoladex
  Arms: Goserelin

SUMMARY:
Menopause increases the risk of metabolic dysfunction-associated steatotic liver disease (MASLD), possibly owing to the abrupt lack of estrogen. Gonadotropin-releasing hormone (GnRH) treatment in endometriosis is regarded as a model of pharmaceutical menopause. Thus, the effect of goserelin acetate, a GnRH analog that results in transient menopause, on hepatic steatosis and fibrosis will be evaluated in this study.

DETAILED DESCRIPTION:
The prevalence of metabolic dysfunction-associated steatotic liver disease (MASLD), which until recently was known as nonalcoholic fatty liver disease (NAFLD), has risen to 30% of the global adult general population, whereas the pharmaceutical interventions against it remain limited. Owing to the epidemiologic and pathophysiologic association of MASLD with obesity, type 2 diabetes mellitus, dyslipidemia and arterial hypertension, the diagnostic criteria for MASLD are similar to those of the metabolic syndrome.

Menopause has been associated with higher MASLD prevalence, with the lack of estrogen being a very plausible pathogenetic contributor to this liver disease. Other pathogenetic contributors of MASLD, including abdominal obesity, increase in insulin resistance (IR) and dysmetabolism of carbohydrates and lipids, are aggravated after menopause, thus adversely contributing to the pathogenesis of MASLD. Regarding the effect of the lack of estrogen on the liver, most to date data are derived from experimental studies, largely showing a favoring effect on MASLD. Epidemiological studies have also shown menopause as an associate of MASLD. However, existing clinical studies are mostly observational, thereby not being able to show a causative association between menopause and MASLD.

Gonadotropin-releasing hormone (GnRH) treatment in disorders such as endometriosis can be regarded as a model of pharmaceutical menopause. More specifically, GnRH analogs, like goserelin acetate, lead to pharmaceutical menopause by suppressing the axis hypothalamus-pituitary-ovaries, thus, causing an iatrogenic, reversible ovarian cessation, which lasts as long as the use of GnRH. The adverse effects of GnRH are generally mild and reversible after their discontinuation.

This is a prospective, interventional non-randomized study, which aims to evaluate the effect of goserelin acetate on hepatic steatosis in women with histologically confirmed endometriosis compared with women with endometriosis that will not receive pharmacological treatment post-surgically.

ELIGIBILITY:
Inclusion Criteria:

* women of reproductive age
* diagnosis of endometriosis. The disease is suspected by patient's individual history (chronic pelvic pain, dyspareunia or/and dysmenorrhea) and the ultrasonographic imaging (chocolate cysts). The diagnosis is confirmed histologically, after laparoscopic surgical treatment and biopsy sampling, which will be interpreted by an independent blinded pathologist.
* use of contraceptives, which is the first line treatment, is contraindicated or the patient does not consent to receive contraceptives, due to personal preferences.
* written informed consent to participate to the study

Exclusion Criteria:

* mean ethanol consumption >10 g/day
* history of other chronic liver disease (e.g., viral hepatitis, autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cholangitis and overlap syndromes, drug-induced liver injury, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency)
* liver cirrhosis
* any malignancy
* chronic kidney disease
* uncontrolled hypothyroidism or hyperthyroidism
* severe sexual hormone disorders (congenital adrenaline hyperplasia, Down syndrome, Turner syndrome).
* use of the following medications within a 12-month period before baseline, which are associated with drug-induced liver injury (DILI): interferon, tamoxifen, amiodarone, aloperidin, glucocorticoids, hormone replacement therapy, contraceptives, anabolic steroids, any medication against tuberculosis, epilepsy or viruses, methotrexate, parenteral nutrition
* use of the following medications within a 12-month period before baseline, which are probably associated with improvement in hepatic steatosis: vitamin E, pioglitazone, insulin, glucagon-like peptide-1 receptor agonists (GLP-1RAs), sodium- glucose co-transporter-2 inhibitors (SGLT-2i), orlistat, ursodeoxycholic acid
* use of any GnRH agonist or antagonist within a 12-month period before baseline

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Hepatic steatosis | 6 months
  Ultrasound-Guided Attenuation Parameter (UGAP) measured on an ultrasound machine GE Logiq E10s.
  Between-within group interactions in UGAP
  UGAP is a non-invasive index based on the attenuation quantification of the ultrasound beam through the hepatic parenchyma, thus used for hepatic steatosis quantification. Cut-off values of ≥ 0.53 dB/cm/MHz, ≥ 0.60 dB/cm/MHz, and ≥ 0.65 dB/cm/MHz have been proposed for the diagnosis of steatosis grade S1, S2, and S3, respectively
Hepatic fibrosis | 6 months
  Liver stiffness (LS) measured with 2D Shear Wave Elastography (2D SWE) on an ultrasound machine GE Logiq E10s.
  Between-within group interactions in LS
  2D SWE is a non-invasive tool measuring the hepatic parenchyma stiffness, thus indirectly suggesting fibrosis stage (F). Cut-offs values of <8.27 kPa, 8.27-9.39 kPa, 9.40-11.88 kPa and ≥11.88 kPa have been proposed for F0-F1, F2, F3, and F4, respectively.

SECONDARY OUTCOMES:
Liver function tests I - ALT and AST | 6 months
  Between-within group interactions will be performed for each of the following parameters:
  Alanine aminotransferase (ALT; IU/l), aspartate aminotransferase (AST; IU/l);
  ALT to AST ratio will be calculated
Liver function tests II - γGT | 6 months
  Between-within group interactions will be performed for:
  γ-glutamyltransferase (GGT; IU/l)
Insulin resistance | 6 months
  Between-within group interactions will be performed for Homeostasis Model Assessment - Insulin Resistance (HOMA-IR), which is calculated by the formula: fasting glucose (mg/dl) × insulin (mU/l)/405, and is an index of insulin resistance; higher score indicates greater insulin resistance.
Lipid profile | 6 months
  Between-within group interactions will be performed for each of the following parameters:
  Total cholesterol (TC; mg/dL) Triglycerides (TG; mg/dL) High-density lipoprotein cholesterol (HDL-C; mg/dL) 4. Low-density lipoprotein cholesterol (LDL-C)
  LDL-C (mg/dL) is calculated by the formula: TC (mg/dl) - HDL-C (mg/dl) - TG (mg/dl)/5.
Non-invasive hepatic steatosis index I - Fatty Liver Index (FLI) | 6 months
  FLI is calculated by the formula [(e0.953 × Loge (TG, mg/dL) + 0.139×BMI (kg/m2) + 0.718× Loge (GGT, U/L) + 0.053 × waist circumference (cm) -15.745) / (1 + e0.953 × Loge (TG, mg/dL) + 0.139×BMI (kg/m2) + 0.718×Loge (GGT, U/L) + 0.053 × waist circumference (cm) -15.745)] × 100.
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis index II - Hepatic Steatosis Index (HSI) | 6 months
  HSI is calculated by the formula: 8 * ALT (U/L) / AST (U/L) + BMI (kg/m2) + 2 [if type 2 diabetes melitus (T2DM)] + 2 (if female).
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis index III - Triglyceride/Glucose Index (TyG) | 6 months
  TyG is calculated by the formula: Ln[TG (mg/dL) * Glu (mg/dL) / 2].
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis index IV - Tyg-BMI | 6 months
  Tyg-BMI is calculated by the formula: TyG * BMI (kg/m2).
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis indices V - NAFLD test | 6 months
  NAFLD test is calculated by the formula: -0.695 + 0.031 * BMI (kg/m2) + 0.003 * TC (mg/dL) + 0.014 * ALT (U/L) + 0.025 * C-reactive protein (CRP) (mg/dL).
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis index VI - Metabolic Score for Insulin Resistance (MetS-IR) | 6 months
  MetS-IR is calculated by the formula: Ln[2 * Glu (mg/dL) + TG (mg/dL)] * BMI (kg/m2) / Ln[HDL-C (mg/dL)].
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis index VII - Lipid Accumulation Product index (LAP) | 6 months
  LAP is calculated by the formula: [WC (cm) - 58] * [TG (mg/dL) / 88.57].
  Between-within group interactions will be performed.
Non-invasive hepatic steatosis index VIII - Liver Fat Score (LFS) | 6 months
  LFS is calculated by the formula: -2.89 + 1.18 (if metabolic syndrome) + 0.45 * 2 (if T2DM) + 0.15 * insulin (mU/L) + 0.04 * AST (U/L) - 0.94 * AST (U/L) / ALT (U/L).
  Between-within group interactions will be performed.
Non-invasive hepatic fibrosis index I - NAFLD fibrosis score (NFS) | 6 months
  NFS is calculated by the formula: -1.675 + 0.037 * age (years) + 0.094 * BMI (kg/m2) + 1.13 (if impaired fasting glucose or T2DM) + 0.99 * AST (U/L) / ALT (U/L) - 0.013 * platelet count [*10(9)/L] - 0.66 * albumin (g/dL).
  Between-within group interactions will be performed.
Non-invasive hepatic fibrosis index II - Fibrosis-4 index (FIB-4) | 6 months
  FIB-4 is calculated by the formula: age (years) * AST (U/L) / {platelet count [*10(9)/L] * √ALT (U/L)}.
  Between-within group interactions will be performed.
Non-invasive hepatic fibrosis index III - AST-to-Platelet Ratio Index (APRI) | 6 months
  APRI is calculated by the formula: AST (U/L) / upper limit of normal * 100 / platelet count [*10(9)/L].
  Between-within group interactions will be performed.
Non-invasive hepatic fibrosis index IV - Metabolic dysfunction-Associated Fibrosis Score (MAF-5) | 6 months
  MAF-5 is calculated by the formula: -11.3674 + 0.0282 * WC (cm) - 0.1761 * BMI (kg/m2) + 0.0019 * WC (cm) * BMI (kg/m2) + 2.0762 (if T2DM) + 2.9207 * Ln[AST (U/L)] - 0.0059 * platelet count [*10(9)/L].
  Between-within group interactions will be performed.
Adiponectin | 6 months
  Adiponectin is measured in μg/mL.
  Between-within group interactions will be performed.
Leptin | 6 months
  Leptin is measured in ng/mL.
  Between-within group interactions will be performed.
Tumor Necrosis Factor-α (TNF-α) | 6 months
  TNF-a is measured in pg/mL.
  Between-within group interactions will be performed.
Sex hormones I - Estradiol | 6 months
  Estradiol is measured in pg/mL.
  Between-within group interactions will be performed.
Sex hormones II - Testosterone | 6 months
  Testosterone is measured in ng/mL.
  Between-within group interactions will be performed.
Sex hormones III - Sex Hormone Binding Globulin (SHBG) | 6 months
  SHBG is measured in nmol/L.
  Between-within group interactions will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios A Anastasilakis, MD, PhDc, Study Director — School of Medicine, Aristotle University of Thessaloniki; Athina I Gkiomisi, MD, PhD, Study Director — 424 General Military Hospital, Thessaloniki, Greece; Dimitrios G Goulis, MD, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki; Angelos Daniilidis, MD, PhD, Study Director — School of Medicine, Aristotle University of Thessaloniki; Athanasios A Anastasilakis, MD, PhD, Study Director — 424 General Military Hospital, Thessaloniki, Greece; Chrysi Nalmpantidou, MD, Study Director — "G. Gennimatas" General Hospital, Thessaloniki, Greece; Stergios A Polyzos, MD, PhD, Principal Investigator — School of Medicine, Aristotle University of Thessaloniki
Locations (2):
- Greece (2):
  - 1st Department of Obstetrics and Gynecology, School of Medicine, Aristotle University of Thessaloniki, Thessaloniki
  - 424 General Military Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researchers upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the publication of the study.
Access Criteria: Yet unknown

REFERENCES:
- [Background] Henry L, Paik J, Younossi ZM. Review article: the epidemiologic burden of non-alcoholic fatty liver disease across the world. Aliment Pharmacol Ther. 2022 Sep;56(6):942-956. doi: 10.1111/apt.17158. Epub 2022 Jul 26. PMID 35880713
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. Hepatology. 2023 Dec 1;78(6):1966-1986. doi: 10.1097/HEP.0000000000000520. Epub 2023 Jun 24. PMID 37363821
- [Background] Alberti KG, Zimmet P, Shaw J. Metabolic syndrome--a new world-wide definition. A Consensus Statement from the International Diabetes Federation. Diabet Med. 2006 May;23(5):469-80. doi: 10.1111/j.1464-5491.2006.01858.x. PMID 16681555
- [Background] Polyzos SA, Lambrinoudaki I, Goulis DG. Menopausal hormone therapy in women with dyslipidemia and nonalcoholic fatty liver disease. Hormones (Athens). 2022 Sep;21(3):375-381. doi: 10.1007/s42000-022-00369-8. Epub 2022 May 9. PMID 35532850
- [Background] Polyzos SA, Goulis DG. Menopause and metabolic dysfunction-associated steatotic liver disease. Maturitas. 2024 Aug;186:108024. doi: 10.1016/j.maturitas.2024.108024. Epub 2024 May 14. PMID 38760254
- [Background] Palmisano BT, Zhu L, Stafford JM. Role of Estrogens in the Regulation of Liver Lipid Metabolism. Adv Exp Med Biol. 2017;1043:227-256. doi: 10.1007/978-3-319-70178-3_12. PMID 29224098
- [Background] Venetsanaki V, Polyzos SA. Menopause and Non-Alcoholic Fatty Liver Disease: A Review Focusing on Therapeutic Perspectives. Curr Vasc Pharmacol. 2019;17(6):546-555. doi: 10.2174/1570161116666180711121949. PMID 29992886
- [Background] Takaesu Y, Nishi H, Kojima J, Sasaki T, Nagamitsu Y, Kato R, Isaka K. Dienogest compared with gonadotropin-releasing hormone agonist after conservative surgery for endometriosis. J Obstet Gynaecol Res. 2016 Sep;42(9):1152-8. doi: 10.1111/jog.13023. Epub 2016 May 26. PMID 27225336
- [Background] Ferrero S, Evangelisti G, Barra F. Current and emerging treatment options for endometriosis. Expert Opin Pharmacother. 2018 Jul;19(10):1109-1125. doi: 10.1080/14656566.2018.1494154. Epub 2018 Jul 5. PMID 29975553
- [Background] DiVasta AD, Laufer MR. The use of gonadotropin releasing hormone analogues in adolescent and young patients with endometriosis. Curr Opin Obstet Gynecol. 2013 Aug;25(4):287-92. doi: 10.1097/GCO.0b013e32836343eb. PMID 23770813
- [Background] Polyzos SA, Kang ES, Boutari C, Rhee EJ, Mantzoros CS. Current and emerging pharmacological options for the treatment of nonalcoholic steatohepatitis. Metabolism. 2020 Oct;111S:154203. doi: 10.1016/j.metabol.2020.154203. Epub 2020 Mar 6. PMID 32151660
- [Background] Polyzos SA, Kountouras J, Tsatsoulis A, Zafeiriadou E, Katsiki E, Patsiaoura K, Zavos C, Anastasiadou VV, Slavakis A. Sex steroids and sex hormone-binding globulin in postmenopausal women with nonalcoholic fatty liver disease. Hormones (Athens). 2013 Jul-Sep;12(3):405-16. doi: 10.1007/BF03401306. PMID 24121382
- [Background] Pafili K, Paschou SA, Armeni E, Polyzos SA, Goulis DG, Lambrinoudaki I. Non-alcoholic fatty liver disease through the female lifespan: the role of sex hormones. J Endocrinol Invest. 2022 Sep;45(9):1609-1623. doi: 10.1007/s40618-022-01766-x. Epub 2022 Mar 18. PMID 35303270